CLINICAL TRIAL: NCT05816915
Title: Complex Lifestyle Modification in the Treatment of Non-alcoholic Fatty Liver Disease
Brief Title: Lifestyle Modification in the Treatment of NAFLD.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Radan Bruha, Head of 4th Internal clinic, General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU23-01-00288
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: NAFLD
Keywords: NAFLD; Cognitive behavioral therapy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Patients with NAFLD and metabolic syndrome will be randomly assigned to a standard care or a professional lifestyle modification counselling during a 1-yr follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional lifestyle modification counselling (behavioral therapy) (Experimental): Lifestyle intervention will be based on CBT (cognitive behavioral therapy) and mindfulness, especially mindful eating by professional organisation STOB.
  Interventions: Behavioral: Cognitive behavioral therapy
- standard care (No Intervention): Patients will have standard care with regular visits at an outpatient Department of Hepatology. Standard recommendations of lifestyle change and weight reduction will be given by hepatologists.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Subjects will receive professional lifestyle intervention conducted by STOB organization. Using CBT and the so-called third wave of CBT, especially mindfulness, the patients will be guided by certified experts to increase motivation and to change eating and exercise habits, which will be mapped before and after the intervention.
  Arms: Professional lifestyle modification counselling (behavioral therapy)

SUMMARY:
The project will study the impact of individually tailored lifestyle counselling compared to standard care on the parameters of NAFLD/NASH in patients with metabolic syndrome. The factors affecting the outcome (including clinical and laboratory parameters and microbiome profiling) will be evaluated.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD), the hepatic manifestation of a metabolic syndrome, is a leading cause of chronic liver disease worldwide. NAFLD is associated with type 2 diabetes, obesity and genetic factors. Despite intensive effort and numerous trials, as of today there is no approved treatment for NAFLD. Weight reduction is recommended, but no long-term control study assessing the evolution of NAFLD/NASH (non-alcoholic steatohepatitis) during lifestyle modification is available.

The main objective of presented project is to compare the progression of NAFLD/NASH in patients with metabolic syndrome randomly assigned to a standard care or a professional lifestyle modification counselling during a 1-yr follow-up. The investigators hypothesize that professionally tailored life-style counselling in patient with metabolic syndrome and NAFLD will improve liver fat content and other non-invasive parameters of liver disease, and factors (including gut microbiota) affecting progression/regression of NAFLD will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with NAFLD and metabolic syndrome

Exclusion Criteria:

* Etiology of liver disease other than NAFLD.
* Presence of malignant disease.
* Uncontrolled cardiovascular disease
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The effect of CBT on liver fat content | 12 months
  The effect of CBT on liver fat content measured by MRS (percentual change from baseline).
The effect of CBT on inflammatory parameters | 12 months
  The effect of CBT on inflammatory biochemical parameters (percentual change from baseline).
The effect of CBT on liver fibrosis | 12 months
  The effect of CBT on liver fibrosis measured by elastography (percentual change from baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Radan Bruha, Prof., Principal Investigator — General University Hospital, Prague
Locations (1):
- General University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized laboratory results.

REFERENCES:
- [Background] Zelber-Sagi S, Ratziu V, Oren R. Nutrition and physical activity in NAFLD: an overview of the epidemiological evidence. World J Gastroenterol. 2011 Aug 7;17(29):3377-89. doi: 10.3748/wjg.v17.i29.3377. PMID 21876630
- [Background] Smid V, Dvorak K, Sedivy P, Kosek V, Lenicek M, Dezortova M, Hajslova J, Hajek M, Vitek L, Bechynska K, Bruha R. Effect of Omega-3 Polyunsaturated Fatty Acids on Lipid Metabolism in Patients With Metabolic Syndrome and NAFLD. Hepatol Commun. 2022 Jun;6(6):1336-1349. doi: 10.1002/hep4.1906. Epub 2022 Feb 11. PMID 35147302
- [Background] Fernandez T, Vinuela M, Vidal C, Barrera F. Lifestyle changes in patients with non-alcoholic fatty liver disease: A systematic review and meta-analysis. PLoS One. 2022 Feb 17;17(2):e0263931. doi: 10.1371/journal.pone.0263931. eCollection 2022. PMID 35176096